CLINICAL TRIAL: NCT03638739
Title: Exercise and Brain Health in Multiple Sclerosis: A Pilot Study
Brief Title: Exercise and Brain Health in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RG-1707-28348
Record Dates: First submitted 2018-08-02; First posted 2018-08-20 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will engage in supervised, twice-weekly exercise following the Physical Activity Guidelines for Adults with MS for 12 weeks at McMaster University. Following this, they will return to their normal daily activities for a further 12 weeks.
  Interventions: Other: Twice-weekly exercise
- Wait-list Control (Experimental): Participants will engage in their usual daily activities for the first 12 weeks of the study, then will engage in supervised, twice-weekly exercise following the Physical Activity Guidelines for Adults with MS at McMaster University for the 2nd 12 weeks.
  Interventions: Other: Twice-weekly exercise

INTERVENTIONS:
Other: Twice-weekly exercise — An individualized exercise plan, incorporating aerobic and resistance exercises, following the Physical Activity Guideline recommendations will be provided for each participant.

SUMMARY:
Physical activity is now recognized as a therapy for Multiple Sclerosis (MS) that not only improves physical fitness and functional mobility, but there is some evidence that it may also positively influence the more invisible symptoms of the disease that represent "brain health" - fatigue, depression and cognitive impairment. One important feature of physical activity is that it reduces inflammation throughout the body and the brain. The goal of this research is to determine whether people with MS feel less fatigue, depression and cognitive impairment after a program of exercise because there is a decrease in the state of inflammation in the brain.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, degenerative disease of the central nervous system, characterized by inflammatory demyelination and axonal degeneration. MS affects approximately 1 in 500 Canadians. There is no cure for MS and the heterogeneous symptoms of the disease makes it difficult to prescribe effective treatment strategies for disease management. While the progression, severity and specific symptom profile vary from person to person, there are three key symptoms associated with brain health- fatigue, depression and cognitive impairment- that invariably lead to poor quality of life and increased health care costs. Unfortunately, the majority of people with MS suffer from these symptoms (fatigue affects ~90%, depression affects ~50% and cognitive impairment affects 40-65%) and a critical challenge with MS is that these symptoms do not present individually. For example, persons with MS who experience depression are more likely to also experience fatigue and/or cognitive impairment, which together may be more detrimental to quality of life than each symptom alone.

New evidence suggests that the three symptoms affecting brain health may be interrelated through a common mechanism of inflammation. Further, physical exercise is known to reduce inflammation and thus is a prime candidate for a novel therapeutic approach to symptom management through its effect on modulating the inflammatory response. Indeed, physical activity is already used to improve the physical status of individuals with MS and evidence-based physical activity guidelines (PAGs) for MS have been developed to guide prescription. However, the guidelines have not been tested for their effects on reducing inflammation and brain health disease systems. Therefore, the proposed research will be the first to evaluate the clinical utility of the PAGs for MS in reducing brain health disease symptoms and improving quality of life, and the first to comprehensively determine the putative effects of inflammation on these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsing-Remitting MS (RRMS) with mild-moderate disability (EDSS 2-5)
* Aged 18-60
* Score of ≥ 10 on MFIS-5*
* Medical clearance to participate in physical activity * The MFIS-5 is an abbreviated version of the 21-item MFIS, consisting of 5 of the 21 items of the MFIS that most strongly correlate with the total MFIS score. A score ≥ 10 on the MFIS-5 is considered to indicate "high-level" of fatigue

Exclusion Criteria:

* Current participation in regular physical activity (at least twice-weekly)
* Other serious medical condition that might impair ability to participate in strength or aerobic exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Fatigue | Outcome will be measured at Baseline, 12 weeks and 24 weeks.
  Changes in perceived fatigue as a result of the intervention will be assessed through changes in scores on the Modified Fatigue Impact Scale (MFIS-21).
Change in Inflammatory Markers | Outcome will be measured at Baseline, 12 weeks and 24 weeks.
  Inflammatory markers will be measured from the blood. Participants will have 15ml of blood drawn by a trained phlebotomist. Levels of serum cytokines (TNF, IL6, IL10, IL1RA) will be measured in using the custom created Milliplex MAP Human Magnetic Bead Panel (Millipore, ON, CA). Cellular immunophenotyping will be performed to test whether there are changes in cellular inflammation.
Change in Depression | Outcome will be measured at Baseline, 12 weeks and 24 weeks.
  Change in depression will be measured with the Hospital Anxiety and Depression Scale (HADS).
Change in Cognition | Outcome will be measured at Baseline, 12 weeks and 24 weeks.
  Changes in cognitive ability will be assessed by using the Brief International Cognitive Assessment for MS (BICAMS) test battery.

SECONDARY OUTCOMES:
Change in Aerobic Capacity | Outcomes will be measured at Baseline, 12 weeks and 24 weeks.
  Participants will perform a progressive exercise test on the cycle ergometer to determine peak oxygen consumption (aerobic capacity). Expired gas and ventilatory parameters will be acquired throughout the protocol using a metabolic cart allowing for the determination of submaximal and maximal oxygen consumption.
Change in Muscle Strength | Outcomes will be measured at Baseline, 12 weeks and 24 weeks.
  The maximum weight that can be lifted in one repetition (1RM) will be assessed in major muscle groups of the upper and lower body to assess muscle strength.
Change in Perceived Quality of Life (QOL) | Outcomes will be measured at Baseline, 12 weeks and 24 weeks.
  Health-related quality of life will be assessed by the disease-specific MS Quality of Life-54 (MSQoL-54) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Activity Centre for Excellence, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No